CLINICAL TRIAL: NCT00379691
Title: Phenylephrine Dose-Finding Study to Minimize Hypotension Due to Spinal Anesthesia for Cesarean Section
Brief Title: Ideal Dose of Phenylephrine to Treat Low Blood Pressure During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 06-01; 06-0186-E
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Last update posted 2007-03-21 (Estimated); Status verified 2007-03

CONDITIONS: Hypotension; Nausea
Keywords: spinal; Cesarean section; hypotension; nausea; vomiting; phenylephrine
MeSH Terms: conditions — Hypotension; Nausea; Vomiting | interventions — Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: phenylephrine

SUMMARY:
The purpose of this study is to determine the minimum effective bolus dose of phenylephrine to prevent post-spinal hypotension in Cesarean section in 95 % of our patients. An adequate response will be defined as the absence of hypotension or nausea/vomiting during the period from induction of spinal anesthesia to uterine incision prior to fetal delivery.

DETAILED DESCRIPTION:
The purpose of this study is to determine the minimum effective bolus dose of phenylephrine to prevent post-spinal hypotension in CS in 95 % of our patients. The study will be conducted in a randomized double-blinded fashion. This dose-response study will be conducted as per the up-down sequential allocation method, modified by the Narayana rule, designed to cluster the results around the ED95.

Blood pressure will be monitored every minute from intrathecal injection to the delivery of the child. Phenylephrine will be administered every time the blood pressure is equal to or lower than the control value.Hypotension will be defined as a SBP less than 80 % of the baseline value, in which case the treatment will be a failure. Hypertension will be defined as a SBP more than 120 % of baseline value. If a patient presents hypertension for two consecutive measurements, the case will be considered a drop out.An adequate response will be defined as the absence of hypotension or nausea/vomiting during the period from induction of spinal anesthesia to uterine incision prior to fetal delivery.

The results of this study will define the minimum effective dose of phenylephrine to prevent post-spinal hypotension and nausea/vomiting secondary to hypotension in Cesarean section, thus optimizing the safety profile with respect to maternal and fetal side effects of this vasopressor.

ELIGIBILITY:
Inclusion Criteria:

* Elective CS under spinal anesthesia
* Normal singleton pregnancy beyond 36 weeks gestation
* ASA physical status I/II
* Weight 50-100 kg, height 150-180 cm
* Age over 18 years

Exclusion Criteria:

* Patient refusal
* Allergy or hypersensitivity to phenylephrine
* Preexisting or pregnancy-induced hypertension
* Cardiovascular or cerebrovascular disease
* Fetal abnormalities
* History of diabetes, excluding gestational diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-08; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the minimum dose of phenylephrine which effectively prevents both hypotension and nausea/vomiting between intrathecal injection of the local anesthetic and delivery of the fetus.

SECONDARY OUTCOMES:
Maternal Demographics: Maternal age-weight-height
Nausea and Vomiting
Time of intrathecal injection, skin incision, uterine incision, and delivery
Total dose of phenylephrine
Hypertension (> 120 % of baseline)
Bradycardia (< 50 bpm)
Upper sensory level of anesthesia by pinprick upon delivery
Umbilical artery and vein blood gases

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD PhD, Principal Investigator — Department of Anesthesia and Pain Management, Mount Sinai Hospital, University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada